CLINICAL TRIAL: NCT00123565
Title: A Randomized Dose Ranging Study of Hexadecasaccharide Including Active Control, in Patients With Unstable Angina or Non-ST-Segment Elevation Myocardial Infarction Scheduled to Undergo Percutaneous Coronary Intervention (SHINE)
Brief Title: Hexadecasaccharide (SR123781A) in Patients With Unstable Angina or Non-ST-Segment Elevation Myocardial Infarction
Acronym: SHINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI5228; SR123781A
Record Dates: First submitted 2005-07-22; First posted 2005-07-25 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Atherosclerosis
Keywords: Coronary Disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease | interventions — SR 123781A

INTERVENTIONS:
Drug: Hexadecasaccharide (SR123781A)

SUMMARY:
The purpose of this study is to test whether SR123781A is a possible treatment for patients with acute coronary syndromes (heart attack) who are scheduled to undergo a percutaneous coronary intervention (PCI) within 48 hours after inclusion in the study. Two doses of SR123781A are currently tested, each in a group of about 180 patients per group to find which is the most adequate, versus heparin and glycoprotein IIbIIIa (GPIIBIIIA) antagonist.

ELIGIBILITY:
Inclusion Criteria:

* A person with a diagnosis of acute coronary syndrome who is scheduled to undergo a PCI within 48 hours.
* A person who is of the legal age of 21, who is mentally competent, and who has signed a written informed consent

Exclusion Criteria:

* A person with known allergy or any contra-indication to active control.
* A person who has received heparin during more than 48 hours before inclusion in the study.
* A person treated with warfarin (oral anticoagulant).
* A person with current bleeding or recognized increased risk of bleeding or history of intracranial hemorrhage.
* A person who has had a stroke within the last 6 months.
* A person with uncontrolled hypertension despite antihypertensive therapy.
* A person with history of clinically significant reduction in blood platelets or neutrophils (white blood cells).
* A person who has laboratory evidence of significantly reduced renal function or who is dependent on renal dialysis.
* A person who has a coronary bypass performed during the previous month.
* A pregnant or nursing woman or a woman of childbearing potential (before menopause) who does not have a negative pregnancy test and does not use a reliable method of birth control.
* A person who has received any investigational treatment in the preceding month.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1257 (Actual)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Efficacy: composite of all causes of death, new myocardial infarction, or severe myocardial ischemia requiring urgent repeat target vessel revascularization within 7 days following randomization.

SECONDARY OUTCOMES:
Safety: Major bleeding according to the criteria of Thrombolysis In Myocardial Infarction study group.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (18):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Buenos Aires, Argentina
- Sanofi-Aventis, Macquarie Park, Australia
- Sanofi-Aventis, Diegem, Belgium
- Sanofi-Aventis, São Paulo, Brazil
- Sanofi-Aventis, Laval, Quebec, Canada
- Sanofi-Aventis, Providencia, Santiago Metropolitan, Chile
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis France, Paris, France
- Sanofi-Aventis, India, India
- Sanofi-Aventis, México, Mexico
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-Aventis, Porto Salvo, Portugal
- Sanofi-Aventis, Moscow, Russia
- Sanofi-Aventis, Seoul, South Korea
- Sanofi-aventis, Barcelona, Spain
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com